CLINICAL TRIAL: NCT00711646
Title: A Double Blind, Randomised, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Cannabis Based Medicine 1:1 THC:CBD Compared With Placebo for the Treatment of Spasticity in Patients With Multiple Sclerosis.
Brief Title: A Study of Sativex® for Relief of Spasticity in Subjects With Multiple Sclerosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWMS0106
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Spasticity; Multiple Sclerosis
Keywords: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental)
  Interventions: Drug: Sativex®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex® — containing THC (27 mg/ml):CBD (25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Maximum permitted dose was eight actuations in any three hour period and 24 actuations (THC 65 mg: CBD 60 mg) in 24 hours
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — containing peppermint oil, 0.05% (v/v), quinoline yellow, 0.005% (w/v), sunset yellow, 0.0025% (w/v), in ethanol:propylene glycol (50:50) excipient.
  Other Names: GW-4001-01
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of Sativex® in subjects diagnosed with MS and spasticity.

DETAILED DESCRIPTION:
This was an eight week (two weeks baseline, six weeks treatment), multicentre, double blind, randomised, placebo controlled parallel group study to evaluate the efficacy, safety and tolerability of Sativex® in subjects diagnosed with MS and spasticity. Subjects were screened to determine eligibility and completed a two week baseline period. Subjects then returned to the site for assessment, randomisation and dose introduction. Visits occurred at the end of treatment week two and at the end of the study (treatment week six) or withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female, aged 18 years or above.
* Stable disease for at least three months prior to study entry, in the opinion of the investigator.
* Diagnosed with MS whose spasticity was not wholly relieved with the therapy at the time of study entry.
* Significant spasticity in at least two muscle groups defined as a score of two or more on the Ashworth Scale for each muscle group.
* Stable dose of current anti-spasticity medication for at least 30 days prior to study entry.
* Willing to maintain a stable dose of anti-spasticity medication and level of physiotherapy for the duration of the study.
* Clinically acceptable laboratory results at Visit 2.
* Willing, if female and of child bearing potential or male subjects with a partner of child bearing potential, to ensure that effective contraception was used during the study and for three months thereafter.
* No cannabinoid use (cannabis, Marinol® or Nabilone) for at least seven days before Visit 1 and were willing to abstain from any use of cannabis during the study.
* Able (in the investigators opinion) and willing to comply with all study requirements.
* Willing for the Home Office to be notified of his or her participation in the study (applicable to the UK centres only).
* Willing to allow his or her GP and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* History of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Known history of alcohol or substance abuse.
* Severe cardiovascular disorder, such as ischaemic heart disease, arrhythmias, poorly controlled hypertension or severe heart failure.
* History of epilepsy.
* Female subject who was pregnant, lactating or planning pregnancy during the course of the study.
* Significant renal or hepatic impairment.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Subject who was terminally ill or was inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the investigator, either put the subject at risk because of participation in the study, or influenced the result of the study, or the subject's ability to participate in the study.
* Regular levodopa (Sinemet®, Sinemet Plus®, Levodopa, L-dopa, Madopar®, Benserazide) therapy within seven days of study entry.
* Male subject receiving sildenafil (Viagra®) and unwilling to stop medication for the duration of the study.
* Subjects who were taking fentanyl (Durogesic®, Actiq®)
* Subjects who were taking antiarrhythmic medications.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medications.
* Known or suspected adverse reaction to cannabinoids.
* Planned travel outside the UK during the study (applicable to the UK centres only).
* Donation of blood during the study.
* Subjects who had participated in another research study in the 12 weeks prior to study entry.
* Subjects previously randomised into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2002-06; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Collin, MB BS MRCP FRCP, Principal Investigator — Royal Berkshire Hospital
Locations (1):
- Royal Berkshire Hospital, Reading, Oxfordshire, United Kingdom

REFERENCES:
- [Result] Collin C, Davies P, Mutiboko IK, Ratcliffe S; Sativex Spasticity in MS Study Group. Randomized controlled trial of cannabis-based medicine in spasticity caused by multiple sclerosis. Eur J Neurol. 2007 Mar;14(3):290-6. doi: 10.1111/j.1468-1331.2006.01639.x. PMID 17355549
- [Derived] Di Marzo V, Centonze D. Placebo effects in a multiple sclerosis spasticity enriched clinical trial with the oromucosal cannabinoid spray (THC/CBD): dimension and possible causes. CNS Neurosci Ther. 2015 Mar;21(3):215-21. doi: 10.1111/cns.12358. Epub 2014 Dec 4. PMID 25475413

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Contains Δ9 tetrahydrocannabinol (THC), 27 mg/ml: cannabidiol (CBD), 25 mg/ml delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose was 48 actuations (THC 130 mg: CBD 120 mg) in 24 hours.
- Placebo: Contains no active drug but colourants and excipients. Maximum permitted dose was 48 actuations in 24 hours.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 124 | 65
Completed | 112 | 62
Not Completed | 12 | 3
Not completed — Adverse Event | 6 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — administrative decision | 0 | 1
Not completed — patient non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 124 | 65 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 118 | 65 | 183
  >=65 years | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (10.2) | 47.8 (9.5) | 49.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 34 | 114
  Male | 44 | 31 | 75
Region of Enrollment [Number; unit: participants]
  United Kingdom | 108 | 56 | 164
  Romania | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change From Baseline in the Mean Spasticity 0-10 Numerical Rating Scale Score.
Description: The spasticity Numerical Rating Scale was completed at the same time each day, i.e. bedtime in the evening. The patient was asked "on a scale of '0 to 10', please indicate the number that best describes your average spasticity in the last 24 hours" where 0 = no spasticity and 10 = worst ever spasticity. For the analysis, end of treatment was defined as the mean of the last seven days in the study or the last three days if the subject withdrew due to worsening spasticity or lack of efficacy. A negative value indicates an improvement in spasticity score from baseline.
Time Frame: 0-52 days
Population: All randomised subjects who received at least one dose of study medication and had on-treatment efficacy data were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 120 | 64
units on a scale | -1.18 (1.83) | -0.63 (1.62)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in mean 11-point Numerical Rating Scale spasticity score was compared between treatment groups using analysis of covariance (ANCOVA). The model included treatment and centre as factors and baseline 11-point Numerical Rating Scale spasticity score as a covariate; Test type: Superiority or Other; p = 0.048, ANCOVA; Estimated mean treatment difference = -0.517, 95% CI 2-sided [-1.029 to -0.004]

2. Secondary Outcome: Change From Baseline in Mean Ashworth Scale Score at the End of Treatment
Description: The mean Ashworth Scale score across muscle groups was calculated using only those muscle groups with a score of greater than or equal to two at baseline. All 20 muscle groups were assessed for spasticity (using a 1-5 scale): 1= no increase in muscle tone to 5= passive movement is difficult and affected part is rigid in flexion or extension. The score for all 20 muscle groups were added to give a total score out of 100; minimum score was 20. A decrease in score indicates an improvement in condition.
Time Frame: Days 0 - 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 114 | 63
units on a scale | -0.64 (0.56) | -0.53 (0.58)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in mean Ashworth Scale score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline Ashworth Scale score as a covariate; Test type: Superiority or Other; p = 0.218, ANCOVA; Estimated mean treatment difference = -0.11, 95% CI 2-sided [-0.29 to 0.07]

3. Secondary Outcome: Change From Baseline in Mean Spasm Frequency Score at the End of Treatment
Description: Each day subjects recorded in their diary the frequency of their spasms using the following scoring system: 0 = no spasms, 1 = one or fewer spasms per day, 2 = between one and five spasms per day, 3 = six to nine spasms per day, 4 = ten or more spasms per day or continuous contraction. For the analysis, end of treatment was defined as the mean of the last seven days in the study or the last three days if the subject withdrew due to worsening spasticity or lack of efficacy.
Time Frame: Days 0 - 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 120 | 64
units on a scale | -0.37 (0.77) | -0.26 (0.74)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in mean spasm frequency score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline spasm frequency score as a covariate; Test type: Superiority or Other; p = 0.141, ANCOVA; Estimated mean treatment difference = -0.17, 95% CI 2-sided [-0.39 to 0.06]

4. Secondary Outcome: Change From Baseline in Mean Motricity Index Score for the Arms
Description: Arm - 3 movements were pinch grip, elbow flexion and shoulder abduction. The total arm score was the addition of the score for the 3 arm movements. One point was then added to give a maximum score of 100; minimum was 1 point. Where both arms were assessed, the average of the two limbs scores was used as the assessment score; otherwise the affected limb total score was used. An increase in score indicates an improvement in condition..
Time Frame: Day 7 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 25 | 15
units on a scale | 3.64 (14.82) | 3.07 (10.08)
Statistical Analysis 1: Comparison: Sativex vs Placebo; The change in mean Motricity Index score was compared between treatment groups using ANCOVA. The model included treatment and centre as factors and baseline Motricity Index score as a covariate; Test type: Superiority or Other; p = 0.766, ANCOVA; Estimated mean treatment difference = 1.30, 95% CI 2-sided [-7.47 to 10.07]

5. Secondary Outcome: Patient's Global Impression of Change in Condition at the End of Treatment
Description: A 7-point Likert-type scale was used, with the question: 'Please assess the change in your condition since entry into the study using the scale below' with the markers "very much improved, much improved, slightly improved, no change, slightly worse, much worse or very much worse". At Visit 2 (Baseline) patients wrote a brief description of their condition which was used at end of treatment to aid their memory regarding their symptoms at study start. For each of above markers the number of participants were reported.
Time Frame: Day 52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 124 | 65
participants
  Very Much Improved | 2 | 0
  Much Improved | 24 | 11
  Minimally Improved | 40 | 20
  No Change | 38 | 26
  Minimally worse | 10 | 5
  Much Worse | 2 | 2
  Very Much Worse | 0 | 0
  Missing | 8 | 1
Statistical Analysis 1: Comparison: Sativex vs Placebo; The proportion of subjects who considered their condition 'Very Much Improved', 'Much Improved' or 'Minimally Improved' was compared between treatment groups using Fisher's Exact Test; Test type: Superiority or Other; p = 0.349, Fisher Exact; Estimated mean treatment difference = 8.46, 95% CI 2-sided [-6.74 to 23.66]

6. Secondary Outcome: Incidence of Adverse Events as a Measure of Subject Safety
Description: The number of subjects who reported an adverse event during the course of the study is presented.
Time Frame: Day 0-52
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 124 | 65
participants | 102 | 46

7. Secondary Outcome: Change From Baseline in Mean Motricity Index Score for the Legs
Description: Ankle dorsiflexion, knee extension and hip flexion were assessed and scored to give a maximum of 100%. The Motricity Index score (scale 1-100) was recorded for limbs that had an associated Ashworth Scale score, which was greater than or equal to two at baseline.
Time Frame: Day 7 and Day 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 103 | 56
units on a scale | 6.01 (12.30) | 2.15 (13.41)
Statistical Analysis 1: Comparison: Sativex vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.054, ANCOVA; Estimated mean treatment difference = 3.86, 95% CI 2-sided [-0.06 to 7.78]

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the time of consent to post study follow up (9 - 10 weeks) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 4/124 | 3/65
Other Adverse Events (participants affected / at risk) | 102/124 | 46/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=124) | Placebo (N=65)
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1
Mobility Decreased (General disorders) | 1 | 0
Bartholin's Abscess (Infections and infestations) | 1 | 0
Urinary Tract Infection NOS (Infections and infestations) | 2 | 1
Lower Respiratory Tract Infection NOS (Infections and infestations) | 0 | 1
Pancreatic Carcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary Incontinence Aggravated (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=124) | Placebo (N=65)
Dizziness (Nervous system disorders) | 40 | 7
Fatigue (General disorders) | 13 | 4
Urinary Tract Infection NOS (Infections and infestations) | 13 | 6
Dry Mouth (Gastrointestinal disorders) | 11 | 4
Balance Impaired NOS (Nervous system disorders) | 9 | 1
Nausea (Gastrointestinal disorders) | 9 | 4
Headache NOS (Nervous system disorders) | 8 | 4
Diarrhoea NOS (Gastrointestinal disorders) | 7 | 2
Oral Pain (Gastrointestinal disorders) | 6 | 7
Somnolence (Nervous system disorders) | 6 | 1
Confusion (Psychiatric disorders) | 6 | 2
Depressed Mood (Psychiatric disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 5 | 1
Disorientation (Psychiatric disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 5 | 1
Disturbance in Attention (Nervous system disorders) | 4 | 0
Euphoric mood (Psychiatric disorders) | 4 | 2
Vision Blurred (Eye disorders) | 4 | 0
Weakness (General disorders) | 4 | 1
Pain in Limb (Musculoskeletal and connective tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.